CLINICAL TRIAL: NCT03879057
Title: Phase I Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Surufatinib Combined With JS001 in Patients With Advanced Solid Tumors
Brief Title: Trial of Surufatinib Combined With JS001 in the Treatment of Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGOG-3006/2018-012-00CH2
Record Dates: First submitted 2018-12-28; First posted 2019-03-18 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib 200mg/JS001 240mg (Experimental): Surufatinib at a dose of 200mg Qd, with humanized anti-PD-1 monoclonal antibody（JS001） injected intravenously 240mg per 3 weeks until disease progresses or unacceptable tolerability occurs.
  Interventions: Drug: Surufatinib/humanized anti-PD-1 monoclonal antibody
- Surufatinib 300mg/JS001 240mg (Experimental): Surufatinib at a dose of 300mg Qd, with humanized anti-PD-1 monoclonal antibody（JS001) injected intravenously 240mg per 3 weeks until disease progresses or unacceptable tolerability occurs.
  Interventions: Drug: Surufatinib/humanized anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Surufatinib/humanized anti-PD-1 monoclonal antibody — humanized anti-PD-1 monoclonal antibody(JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with th combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activitation of lymphocytes and elimination of malignancy theoretically.
  Other Names: Surufatinib/JS001

SUMMARY:
This is an open-label, phase I study evaluating safety, tolerability, pharmacokinetics and efficacy of Surufatinib combined with the humanized anti-PD-1 antibody JS001 in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
2. Male and Female aged between 18 and 75 years are eligible;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
4. Histologic diagnosis of locally advanced or metastatic unresectable solid tumors (neuroendocrine tumors, liver carcinoma, gastric carcinomas considered with priority);
5. Failed after standard treatment (disease progression or intolerable for toxic side effects) or no effective to treatment;
6. For liver carcinoma with Child-Pugh of grade A and grade B (≤ 7 points);
7. Radiographic evidence of disease rogression by RECIST criteria on or after last anti-cancer therapy within 6 months; If the single lesion previously received radiation, ablation, there must be an imaging identification for disease progression;
8. Predicted survival >=3 months;
9. At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
10. Screening laboratory values must meet the following criteria (within past 14 days): hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN, creatinine clearance >50ml/min (CockcroftGault equation) PT/INR, aPTT≤1.5 x ULN;
11. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.

Exclusion Criteria:

1. The toxicity associated with previous anti-tumor treatment has not recovered to ≤CTCAE1, except for peripheral neurotoxicity and alopecia ≤CTCAE2 caused by oxaliplatin;
2. Had other malignant tumors in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled);
3. Evidence with active CNS disease;
4. Prior treatment with chemotherapy, biological immunotherapy, targeted therapy, Chinese herbal medicine within 2 weeks.
5. Prior treatment with radical radiation within 4 weeks
6. Prior treatment with antiPD1/PDL1/PDL2/CTLA-4 antibody or Sulfatinib;
7. Prior treatment with corticosteroids (dose > 10 mg/day prednisone or other hormones) or other immunosuppressive agents within 2 weeks, nasal or inhalation in allowed (dose > 10 mg/day prednisone or other hormones).
8. Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
9. Prior live vaccine therapy within past 4 weeks;
10. Prior major surgery within past 4 weeks (diagnostic surgery excluded);
11. Uncontrolled malignant pleural effusion, ascites or pericardial effusion;
12. Hypertension that is not controlled by the drug, and is defined as: SBP≥140 mmHg and/or DBP≥90 mmHg;
13. The patient currently has disease or condition that affects the absorption of the drug, or the patient cannot be administered orally;
14. Received a potent inducer or inhibitor of CYP3A4 within 2 weeks, or continue receiving these drugs during the study;
15. Digestive tract disease such as gastric and duodenal active ulcer, ulcerative colitis or unresected tumor, or other conditions determined by the investigator that may cause gastrointestinal bleeding and perforation;
16. Evidence of bleeding tendency or history within 2 months, or thromboembolic event (including a stroke event and/or a transient ischemic attack) occurred within 12 month;
17. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, LVEF <50%, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
18. Clinically significant severe electrolyte abnormality judged by investigator ;
19. Active infection or unexplained fever during the screening period (temperature >38.5C)
20. History with tuberculosis who are receiving or have received anti-TB treatment within 1 year.
21. Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia, severe impaired lung function, etc; Radiation pneumonitis in the radiotherapy area is allowed;
22. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>2000IU/ml);
23. Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
24. Pregnant or nursing;
25. Hypersensitivity to Sulfatinib or recombinant humanized antiPD1 monoclonal Ab;
26. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
adverse events | 1 year
  Safety of participants followed for the duration of hospital stay, an expected average of 1 week
Maximum tolerated dose | 4 week
  tolerability during the treatment of first cycle

SECONDARY OUTCOMES:
Objective response rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation. CT/MRI will be performed every 2 cycles of treatment by RECIST 1.1(each cycle is 21 days))
time to treatment failure(TTF) | 1 month
  From date of enrollment until the date of tumor progression
Maximum Plasma Concentration (Cmax) | 8 days
  Pharmacokinetic profile in terms of observed maximum plasma concentration
Area Under the Curve From Time Zero Extrapolated to Infinity (AUC(0-inf)) | 8 days
  Pharmacokinetic profile in terms of plasma concentration-time curve from time zero extrapolated to infinity, AUC(0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, PhD, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Lu M, Sun Y, Gong J, Li J, Lu Z, Li J, Zhang X, Li Y, Peng Z, Zhou J, Wang X, Shen L. Surufatinib plus toripalimab in patients with advanced solid tumors: a single-arm, open-label, phase 1 trial. J Cancer Res Clin Oncol. 2023 Feb;149(2):779-789. doi: 10.1007/s00432-021-03898-8. Epub 2022 Feb 15. PMID 35166929